CLINICAL TRIAL: NCT01963325
Title: Phase II Study of Abraxane Plus S-1 as Second-line Treatment for Cholangiocarcinoma
Brief Title: S-1 in Combination With Abraxane in Treating Cholangiocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yuhong Li (Other)
Responsible Party: Sponsor-Investigator, Yuhong Li, MD, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S1vsNab-P20130819
Record Dates: First submitted 2013-09-26; First posted 2013-10-16 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — S 1 (combination); Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- S-1 plus Abraxane (Experimental): Patients will receive Abraxane at 100 mg/m2 X 3 doses on Days 1, 8. S-1 chemotherapy was given based on the body surface area, <1.25 m2: 80mg/day, 1.25~1.5 m2: 100mg/day, ≧1.5 m2: 120mg/day. Given orally twice daily for 14 days, followed by 7 days without treatment.
  Interventions: Drug: S-1 plus Abraxane

INTERVENTIONS:
Drug: S-1 plus Abraxane — Patients will receive Abraxane at 100 mg/m2 X 3 doses on Days 1, 8. S-1 chemotherapy was given based on the body surface area, <1.25 m2: 80mg/day, 1.25~1.5 m2: 100mg/day, ≧1.5 m2: 120mg/day. Given orally twice daily for 14 days, followed by 7 days without treatment.
  Other Names: Paclitaxel Albumin-Bound Particles for Injectable Suspension; Gimeraciland Oteracil Porassium Capsules

SUMMARY:
This phase II study was designed to evaluate the efficacy and safety of S-1 plus Abraxane as second-line treatment for cholangiocarcinoma.

DETAILED DESCRIPTION:
There are no standard second-line treatment for cholangiocarcinoma, new therapies are needed. The efficacy of S-1 as first-line treatment for cholangiocarcinoma was confirmed in several studies. The IMPACT study showed that Abraxane plus gemcitabine provide better survival than gemcitabine alone. Since cholangiocarcinoma displayed similar sensitivity to chemotherapy which was used in pancreatic carcinoma, we assume that S-1 plus Abraxane is effective and safe in treating cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of cholangiocarcinoma
* Not eligible for curative surgery
* Progressed after first-line gemcitabine-based chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or better
* No serious or uncontrolled concomitant medical illness
* Adequate bone marrow function (absolute neutrophil count ≧1,500 ul, platelet count ≧90,000/ul), hemoglobin: > or equal to 8 mg/dL, total bilirubin: < or equal to 1.5 X institutional upper limit of normal, calculated creatinine clearance greater than or equal to 60 mL/min (calculated by the Cockcroft and Gault method).

Exclusion Criteria:

* Uncontrolled infection or severe active comorbid disease
* Previous malignancy in the past five years, excluding nonmelanoma skin cancers and in situ cervical, bladder or uterine cancer
* Pregnancy or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-08; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Response rates | 6 months

SECONDARY OUTCOMES:
Progression-free survival | 6 months
Number of participants with adverse events | 12 months
  Adverse events evaluated by Common Terminology Criteria for Adverse Events v3.0.

CONTACTS AND LOCATIONS:
Overall Officials: Yuhong Li, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China